CLINICAL TRIAL: NCT04295993
Title: The Effect of Methylene Blue on Microcirculation in Patients With Septic Shock: a Randomized Controlled Trial
Brief Title: Methylene Blue and Microcirculation in Septic Shock
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareman Mohammad Saad Eldin Abd El Ghafar, Assistant lecturer of anesthesia and critical care medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-13-2019
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Methylene Blue; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methylene blue group (Experimental): The patients in this group will receive methylene blue bolus in addition to the norepinephrine infusion.
  Interventions: Drug: Methylene Blue; Drug: Norepinephrine infusion
- Norepinephrine group (Active Comparator): The patients in this group will receive norepinephrine infusion.
  Interventions: Drug: Norepinephrine infusion

INTERVENTIONS:
Drug: Methylene Blue — The patient will receive Methylene Blue bolus with a dose of 2 mg/kg over 10 minutes.
  Arms: methylene blue group
Drug: Norepinephrine infusion — The patient will receive norepinephrine infusion to maintain mean arterial pressure above 65 mmHg
  Other Names: Levophed

SUMMARY:
This trial aims to identify the effects of methylene blue infusion on the the micro-circulation in patients with septic shock. The investigators will evaluate various indices of micro-circulation such as: microvascular ﬂow index, the flow heterogeneity index, the total vessel density, the perfused vessel density, and the proportion of perfused vessels.

DETAILED DESCRIPTION:
The mortality rate of patients with septic shock remains very high. Arterial hypotension, related to arteriolar vasodilation and myocardial depression are the mainstays of septic shock pathology.

At the level of the micro-circulation, there is insufficient delivery of oxygen to organs and tissues which results in organ dysfunction and potential organ necrosis.One key factor leading to vascular dysfunction is the inappropriately increased production of nitric oxide within the blood vessel endothelium. Elevated levels of nitric oxide results in the blood vessel endothelium receiving direct vasodilator input, as well as the inability to respond to norepinephrine-mediated vasoconstriction. Nitric oxide activates the soluble isoform of the enzyme guanylatecyclase, which in turn increases production of cyclic guanosine monophosphate. Nitric oxide has other beneficial effects which are mediated via other pathways than guanylatecyclase; therefore, administration of a guanylate cyclase inhibitor such as methylene blue could be a safer therapeutic option than the inhibition of nitric oxide production.

These effects of methylene blue could be related to vasoconstriction and positive inotropic effects as well to an increase in blood volume, itself related to a decrease in vascular permeability. The use of methylene blue has been recently advocated as a potential adjunct in the treatment of shock states. However, the effect of MB at the level of the capillary bed, where vital exchange of oxygen and nutrients occurs, is unknown. Thus in this study, the investigators will investigate the effect of methylene blue in combination with NE at the microvascular level in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock
* The patient is on norepinephrine infusion

Exclusion Criteria:

* Elevated serum creatinine (above 1.4 mg/dL)
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-03-10 (Estimated); Primary Completion 2020-09-10 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Microvascular flow index | 6 hours
  The image will be divided into four quadrants and the vessels <20 μ m diameter will be assigned a score based on the predominant flow characteristics of the vessels in that quadrant (0 = absent flow; 1 = intermittent; 2 = sluggish; 3 = normal). The values in each quadrant will be averaged to give an microvascular flow index for each sublingual site at each time point. To determine heterogeneity of perfusion, the flow heterogeneity index will be calculated as the highest microvascular flow index minus the lowest microvascular flow index divided by the mean microvascular flow index.

SECONDARY OUTCOMES:
Total vessel density | 6 hours
  The number of vessels per millimeters squared.
Perfused vessel density | 6 hours
  The number of vessels multiplied by the fraction of perfused vessels
Proportion of perfused vessel | 6 hours
  The number of vessels with flows 2 and 3 divided by the total number of vessels and multiplied by 100.
mean arterial pressure | 24 hours
  the mean arterial blood pressure measured in mmHg
serum lactate | 6 hours
  the value of lactate in the serum measured in milligrams per liter
length of stay in the intensive care unit | 28 days
  the duration of stay in the intensive care unit measured in days
cardiac output | 24 hours
  The amount of blood ejected by the heart in one minute measured in liters
total consumption of norepinephrine | 6 hours
  the total consumption of norepinephrine in 6 hours measured in micrograms.
incidence of mortality | 28 days
  The number of dead patients divided by the total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Principal Investigator — Professor of anesthesia
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No